CLINICAL TRIAL: NCT04667364
Title: Modulation of Pain Sensitization in Complex Regional Pain Syndrome
Brief Title: Pain in Complex Regional Pain Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Niels-Peter Brøchner Nielsen, PhD, Principal Investigator, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRPSprojekt
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Complex Regional Pain Syndrome Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group MED (No Intervention): A group of participants that receives treatment as usual that consists of medicinal treatment, prescribed by a specialist doctor (Carsten Kock-Jensen, MD) from the CRPS clinic and will be monitored using patients' medicinal records.
- Group TENS (Experimental): A group of participants that receives transcutaneous electrical nerve stimulation (TENS) which is an inexpensive, noninvasive and safe treatment for pain.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Conventional TENS will be performed using two electrodes placed on the involved extremity and with the following stimulation parameters; a frequency of 100 Hz, pulse duration 50-100 ms, and at an intensity gradually increased until the patient feels a strong, tolerable and non-painful sensation (18, 19). The intensity is incrementally increased based on patient feedback. Patients will receive guidelines on how to use the TENS device at home and will over a period of 30 days self-administer TENS as needed. Patients is to fill out a predefined schedule on paper each day to monitor dose.
  Arms: Group TENS

SUMMARY:
CRPS is a complex pain condition that usually develops in response to trauma and immobilization which is very painful and debilitating. There is no consensus about the underlying mechanisms which might be a combination of mentally and physically factors. At the moment, better diagnostic clarification and better pain relieving treatment is needed. The aim of this study is to investigate changes in the perception of pain in patients with Complex Regional Pain Syndrome (CRPS), and whether this perception can be affected by treatment with transcutaneous electrical nerve stimulation (TENS) on the painful area. The study will consist of two parts. One in which patients' perception of pain will be compared to the perception of pain in healthy controls. Another in which the included patients are randomly allocated into a group receiving medical treatment plus treatment with transcutaneous electrical nerve stimulation on the painful area or in a group receiving medical treatment as usual (MED).Patients will be evaluated four times. At the start of the study, immediately after treatment, and again at 6 and 12 months after treatment. The evaluation consists of an overall assessment of pain, response to standardized sensory stimuli, and questionnaires about quality of life, physical capacity and mentally/socially well-being.

DETAILED DESCRIPTION:
BACKGROUND Chronic pain represents a major challenge worldwide, with significant clinical, social and economic implications. Complex regional pain syndrome (CRPS) is a chronic pain condition that usually, but not exclusively, develops in response to acute trauma or surgery. It is characterized by pain disproportionate to the preceding trauma, in addition to sensory abnormalities and autonomic disturbances, trophic changes and impaired motor function. Reports indicate that the incidence of CRPS is 26.2/100.000 life-years, with a 3.5:1 female male ratio, and with a mean age at diagnosis 52.7y. The condition is complex and is probably the result of multimodal pathogenesis, that has a significant impact on daily functioning and quality of life (QoL). In addition, few cases resolve completely within 12 months of onset, has a large impact on work ability and some develop chronic pain and disability. The socioeconomic consequences are therefore substantial and an increased focus on CRPS diagnosis and treatment is needed. Because of the complexity of the condition, treatment is difficult and include physiotherapy, education, spinal cord stimulation (SCS) and medical treatment. Primary treatment involves medical treatment which might include important adverse effects such as fatigue, insomnia, anxiety and weight gain, to name a few. Regardless, results vary significantly. One explanation is the multimodality of pain that involves both peripheral nerves, the spinal cord and higher brain centers, modulated by immune cells, interneurons, descending pathways, cognitive and psychosocial factors. Changes in pain sensitization has been proposed to be a driving factor in CRPS and is the result of distorted somatosensory signaling in the central nervous system. Pain normally reflects damaging peripheral input, acting as an important protective function, however, this concept might get distorted so that pain no longer represent peripheral noxious stimuli but rather functional changes of the central nervous system. The pain in these situations arises spontaneously, can be elicited by normally innocuous stimuli (allodynia), is exaggerated and prolonged in response to noxious stimuli (hyperalgesia), and spreads beyond the site of injury (secondary hyperalgesia). Testing some of the underlying mechanisms provides the means to directly evaluate these pain symptoms suggested to be among the primary complaints in CPRS. Accordingly, a range of sensory changes has been suggested including thermal and mechanical hyperalgesia and hypoesthesia. A study found hyperalgesia to blunt pressure in patients with CRPS and with peripheral nerve injury, which has been confirmed by others, suggesting an importance of deep somatic structures such as muscles and bones. Another study showed changes in thermal sensitivity with both heat and cold hyperalgesia in the acute phase of CRPS and a modulation of thermal detection thresholds as the CRPS progressed. In addition, a study reported changes in endogenous pain modulation, implying a shift towards facilitation, whereas others found limited change. These differential results alongside heterogeneous mechanisms associated with diverse clinical features complicates treatment significantly which might only affect a small portion of patients. It is crucial to establish whether patients can be identified and distinguished to facilitate optimal decisions and effects of treatment strategies. This project applies a psychophysical method, based on conventional quantitative sensory testing (QST), to quantify somatosensory function in CRPS patients, to provide a mechanisms-based approach to diagnosis and treatment. Recently QST has been used to complement traditional neurological testing, with greater precision and reliability when assessing somatosensory aberrations and its clinical value is well recognized. Nevertheless, because of a lack of standardization and a paucity in normative data, the application of QST in clinical settings remains scarce. The current project applies QST methodology developed at the Spine center of Southern Denmark, Lillebaelt Hospital, specifically designed to meet clinical demands and will be part of a novel initiative to implement and standardize QST in clinical practice in Denmark. The methodology might prove valuable in a range of different pathologies such as headache, fibromyalgia and diabetic neuropathy. In addition, the current project will combine QST measurement with functional measurements and patient reported outcomes on depression, anxiety and sleep using a national database on pain in collaboration with Pain Center South, University Hospital Odense. The modulation of QST, their interaction and time course together with functional measurements and PRO-data might be a powerful combination for the diagnosis of patients, monitoring and prediction of therapy success. A therapy often used as an adjunct to medication is transcutaneous electrical nerve stimulation (TENS) which is an inexpensive, noninvasive and safe treatment for pain. Electrical stimulation is delivered to peripheral sensory nerves using surface electrodes and has been shown to have a beneficial effect on centralized pain, showing normalized hyperalgesia post intervention. Nevertheless, the beneficial effects remain controversial as more high-quality studies are needed. In addition, pain is complex and depends on contextual, social, psychological and biological factors not necessarily attributed to a specific pathology. These are rarely considered concurrently. The current project will evaluate the effect of TENS, in respect to patients psychological, functional and somatosensory profile, adding valuable information to the existing body of literature.

The aim of the current project is three-fold; 1) to test the feasibility and validity of standardized quantitative sensory testing for CRPS in clinical practice, 2) to evaluate changes in sensitization and 3) to evaluate the effectiveness of transcutaneous electrical nerve stimulation (TENS) and identify subgroups that benefit the most.

The investigators hypothesize that quantitative sensory testing is feasible in a clinical setting and will in combination with functional measurements and PRO-data be a valuable tool for the diagnosis of patients and for the monitoring and prediction of therapy success.

TRIAL DESIGN The project will utilize quantitative methods and strong randomized controlled research designs. The project will consist of two parts; 1) Evaluation of CRPS patient compared to healthy controls, and validation of method. Participants will be assessed at baseline prior to treatment with QST (mechanical stimulation, pain thresholds, cold/heat sensitivity) as outcome measure to identify somatosensory profiles of CRPS patients compared to normative data. 2) Evaluation of treatment with TENS compared to treatment as usual. Patients will be randomly allocated to either a TENS intervention group (TENS) or a treatment as usual group (MED) and will be assessed at baseline, re-test pre TENS, post intervention and 3 month post intervention. Outcomes include QST and patient reported outcomes (pain, quality of life, depression, anxiety, sleep, a.m.). Subsequent analysis of data is planned, to evaluate its ability to predict therapeutic outcomes of TENS.

RECRUITMENT AND SAMPLE SIZE Patients will be recruited from the clinic for CRPS and neuropathic pain, Hospital of South West Jutland, (SVS), University Hospital of Southern Denmark. The clinic functions as a specialized CRPS clinic in the Region of Southern Denmark. Healthy controls will be recruited amongst staff at SVS and partners, relatives or friends.

The planned number of trial participants is based on the assumed superiority of TENS treatment over control. Estimating the sample size for a two-sample means test with a level of significance at 0.05, assuming a common standard deviation (SD) of 2 in NRS pain intensity scores indicates that for the intention-to-treat (ITT) population, 34 individuals is required to obtain a power of at least 80% to establish a minimal clinically significant difference (MCSD) of 2 in NRS pain scores. The MCSD and common standard deviation is based on previous findings with a similar patient group and intervention. With an expected drop-out rate of 20%, a total of 46 individuals will be included in the project, 23 in each group.

ALLOCATION All patients will be evaluated at baseline and their QST data will be compared to a group of healthy controls (Part 1). Subsequently, in part 2, patients will be randomized with a computer-generated block randomization with a 1:1 allocation ratio using random block sizes of 2, 4 and 6 in either group TENS or group MED. The randomization restrictions will not be disclosed, and the sequence will be performed by an external party.

INTERVENTIONS TENS. Conventional TENS will be performed using two electrodes placed on the involved extremity and with the following stimulation parameters; a frequency of 100 Hz, pulse duration 50-100 ms, and at an intensity gradually increased until the patient feels a strong, tolerable and non-painful sensation. The intensity is incrementally increased based on patient feedback. Patients will receive guidelines on how to use the TENS device at home and will over a period of 30 days self-administer TENS as needed. Patients is to fill out a predefined schedule on paper each day to monitor dose (see appendix).

Treatment as usual. Consist of medicinal treatment, prescribed by a specialist doctor (Carsten Kock-Jensen, MD) from the CRPS clinic and will be monitored using patients' medicinal records.

STATISTICAL METHODS To evaluate the empirical distributions of the continuous outcomes, visual inspection of the studentized residuals will be applied to evaluate whether the assumption of normality is reasonable. The treatment groups will be examined for comparability based on baseline demographic and prognostic measures. An Intention-To-Treat (ITT) analysis will be used for all allocated patients and a mixed effects model will be used on the continuous outcome measures to determine the effects of TENS treatment from baseline to post treatment and follow-ups [Between groups factor: TENS vs MED, within groups factor: time]. The model will use robust estimation methods to account for outliers. Finally, a multiple imputation approach will be used in case of missing data. All p-values < 0.05 will be considered statistically significant.

ETHICS AND SIGNIFICANCE The project is to be approved by the Regional Committee on Health Research Ethics for Southern Denmark and will be conducted according to the declaration of Helsinki.

The combination of quantitative pain measurements and PRO-data might be a powerful combination for the diagnosis of patients and monitoring and prediction of therapy success. It might have the potential to provide patients with individualized mechanism-based pain therapy and clarify to what extend and to whom TENS is beneficial. This might result in increased functional capacity and quality of life as a result of significant pain relief. This could have a significant impact on patients' lives as well as significant socioeconomic consequences.

ELIGIBILITY:
Inclusion Criteria:

* CRPS according to existing diagnostic criteria
* Numeric Rating Scale (NRS) pain >4

Exclusion Criteria:

* Prior use of TENS for the past 6 months
* Active inflammatory conditions
* Pacemaker
* Comorbid disease that could cause neuropathic pain such as diabetic neuropathy
* Significant cognitive deficits
* Chronic pain syndrome (e.g. fibromyalgia, phantom pain, rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
NRS pain score | Pre- and 1 week post TENS
  Change in the NRS pain score pre- and post TENS treatment compared with the MED group (controls)

SECONDARY OUTCOMES:
Mechanical pressure pain threshold | Pre, retest and 1, 12 weeks post TENS
  Change in the mechanical pain threshold pre- and post TENS treatment compared with the MED
Temporal summation | Pre, retest and 1, 12 weeks post TENS
  Change in the temporal summation pre- and post TENS treatment compared with the MED
Thermal sensitivity | Pre, retest and 1, 12 weeks post TENS
  Change in thermal sensitivity pre- and post TENS treatment compared with the MED
Conditioned pain modulation | Pre, retest and 1, 12 weeks post TENS
  Change in conditioned pain modulation pre- and post TENS treatment compared with the MED
Use of Analgesics | Pre and 1, 12 weeks post TENS
  Change in use of analgesics pre- and post TENS treatment compared with the MED
Number of Adverse effect | Pre, retest and 1, 12 weeks post TENS
  Number and severity of adverse effects.
Quality of Life measured by SF-36 questionnaire | Pre and 1, 12 weeks post TENS
  Change in health related quality (SF36) of life pre- and post TENS treatment compared with the MED
Functional capacity as measured by the Patient Specific Functional Scale | Pre and 1, 12 weeks post TENS
  Change in functional capacity (PSFS) pre- and post TENS treatment compared with the MED
Pain acceptance measured by the Chronic Pain Acceptance Questionnaire (CPAQ) | Pre and 1, 12 weeks post TENS
  Change in pain acceptance pre- and post TENS treatment compared with the MED
Depression as measured by the Patients Health Questionnaire-9 (PHQ-9) | Pre and 1, 12 weeks post TENS
  Change in depression (PHQ9) pre- and post TENS treatment compared with the MED

CONTACTS AND LOCATIONS:
Overall Officials: Bibi (Valgerdur) Gram, PhD, Study Director — Esbjerg Hospital - University Hospital of Southern Denmark; Carsten Kock-Jensen, MD, Study Director — Esbjerg Hospital - University Hospital of Southern Denmark; Niels-Peter B Nielsen, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of Southwest Jutland, Esbjerg, Region Syddanmark, Denmark